CLINICAL TRIAL: NCT04466306
Title: SARS-CoV2 Pediatric Acute Kidney Injury Registry and Collaborative
Brief Title: Pediatric Acute Kidney Injury in COVID-19
Acronym: SPARC-1
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Children's of Alabama (Other); The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Other Study IDs: ChildrensHA
Record Dates: First submitted 2020-06-24; First posted 2020-07-10 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-07

CONDITIONS: Acute Kidney Injury; COVID
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is an observational registry of children with or suspected to have SARS CoV2 (COVID-19) admitted to pediatric intensive care units (PICU). This registry will help describe the prevalence, rate and severity of acute kidney injury (AKI) in children with Severe Acute Respiratory Syndrome Coronavirus-2(SARS CoV2) across the world. The registry will be developed using a point prevalence methodology and then full retrospective review. Once a week, from April through June 2020, data collection will occur in "real-time" to estimate a weekly point prevalence of AKI and renal replacement therapy (RRT). The operational definition of "patients under investigation" (PUIs) will be used to identify the denominator of patients to be studied. The PUIs will be cohorted into SARS CoV2 test positive, test negative, test pending, or test unavailable. The primary aim of this study is to deliver a global, objective data driven analysis of the burden of AKI in virus positive patients or patients under investigation (PUI) who are admitted to the pediatric intensive care unit.

DETAILED DESCRIPTION:
The primary purpose of the data collection will be to provide a descriptive analysis of the burden and characteristics of AKI in children with SARS-CoV2 proven or suspected infection across the world. This is a prospective, point prevalence study. Data collection will occur once a week during the months of April through June 2020.

The protocol for the point prevalence is for each individual participating site to conduct a surveillance study on predetermined dates of their intensive care units (pediatric medical, surgical, cardiac ICUs) for patients by the inclusion and exclusion criteria. The study is strictly observational. Data will only be captured on the predetermined dates listed. The dates have been chosen to reflect the estimated surge and peak of the virus spread in North America, Europe, Africa, Asia, and Australia. The rationale for performing an urgent point prevalence estimation study first, includes the following: a) there is almost no knowledge on AKI rate, severity of AKI or how current pandemic-setting AKI phenotype differs from what we know of AKI in children prior to the pandemic. A rapidly-performed, high feasibility-designed point prevalence estimation study, with minimal data collection will provide rapid, almost instantaneous dissemination of results to the international community. Based on the results of this study, a follow-up study is planned for a full retrospective data collection of all viral positive patients. Understanding the burden of pediatric AKI during this pandemic within the current context of acute health burden in the healthcare settings and enable planning and feasibility evaluation for quality of care measures and potentially for upcoming technology needs and/or sharing of RRT technology with adult care units; b) an urgent point-prevalence estimation study with minimal but key data collection will inform on any changes to design, sample size requirements or data points for the larger granular longitudinal retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* Patient less than or equal to 25 years of age
* Receiving clinical care in the pediatric intensive care unit (PICU) on a study day in April - June 2020
* Patient considered a "Person Under Investigation" and/or tested positive for SARS-CoV2 (COVID-19)

Exclusion Criteria:

• None

Ages: 7 Days to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients admitted to the pediatric medical, surgical, or cardiac ICU for any condition - with a suspicion for or proven diagnosis of SARS-COV2 (COVID-19).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury (AKI) | 14 days
  Kidney Disease Improving Global Outcomes (KDIGO) Staged AKI by serum creatinine or urine output

SECONDARY OUTCOMES:
Survival | 14 days
  Survival to ICU discharge or Day 14
Rate of Extracorporeal Therapy Requirement | 14 days
  The use of extracorporeal membrane oxygenation (ECMO) and/or renal replacement therapy
Fluid overload | Day of Enrollment
  >20% fluid overload as defined as the net fluid balance since ICU admission (in liters) divided by ICU admission weight
Rate of nephrotoxic medication exposure | Day of Enrollment
  The exposure of enrolled patients to known nephrotoxic medications, including diuretics

CONTACTS AND LOCATIONS:
Overall Officials: Rajit K Basu, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (47):
- United States (33):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Arkansas Children's Research Institute, Little Rock, Arkansas
  - Cedars-Sinai Maxine Dunitz Children's Health Center, Los Angeles, California
  - UCLA Mattel Children's Hospital, Los Angeles, California
  - Lucile Packard Children's Hospital Standford, Palo Alto, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale New Haven Children's Hospital, New Haven, Connecticut
  - UF Health Shands Children's Hospital, Gainesville, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Comer Children's Hospital - UChicago Medicine, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - Children's Mercy, Kansas City, Kansas
  - John Hopkins Children's Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Beaumont Children's Hospital, Royal Oak, Michigan
  - St. Louis Children's Hospital of Washington University, St Louis, Missouri
  - Oishei Children's Hospital of Buffalo, Buffalo, New York
  - Golisano Children's Hospital - University of Rochester Medicine, Rochester, New York
  - Stony Brook Children's Hospital, Stony Brook, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Duke Children's Hospital and Health Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Lifespan Hasbro Children's Hospital, Providence, Rhode Island
  - Medical University of South Carolina Shawn Jenkins Children's Hospital, Charleston, South Carolina
  - Seattle Children's Hospital, Seattle, Washington
- Canada (3):
  - Stollery Children's Hospital, Edmonton, Alberta
  - McMaster Children's Hospital, Hamilton, Ontario
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
- Israel (2):
  - Soroka University Medical Center, Beersheba
  - Dana-Dwek Children's Hospital, Tel Aviv
- Shizuoka Children's Hospital, Shizuoka, Japan
- Serbia (2):
  - Institute for Mother and Child Healthcare, Belgrade
  - University Children's Hospital, Belgrade
- Hospital 12 de Octubre, Madrid, Spain
- United Kingdom (5):
  - Birmingham Children's Hospital NHS, Birmingham
  - Alder Hey Children's Hospital NHS, Liverpool
  - King's College Hospital NHS, London
  - St. George's University Hospital NHS, London
  - Great Ormond Street Hospital NHS, London

IPD SHARING:
Plan to Share IPD: No